CLINICAL TRIAL: NCT02163564
Title: Development of an Insomnia Treatment for Depressed Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Deirdre A. Conroy, Clinical Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 501
Record Dates: First submitted 2014-06-06; First posted 2014-06-13 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Insomnia; Depression
Keywords: Adolescent; Depression; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Focus groups (No Intervention): The first part of the study is to conduct focus groups of adolescents with insomnia and depression. The treatment arm is informed by responses provided by teens in the focus group portion.
- Treatment (Active Comparator): A modified cognitive behavioral therapy for insomnia is the treatment intervention in this treatment arm.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — A non-pharmacological therapy for insomnia based on behavior and cognitive therapy approaches
  Other Names: CBTI
  Arms: Treatment

SUMMARY:
Major depressive disorder (MDD) occurs at least 11% of adolescents and approximately 53-90% of those adolescents have insomnia. If left untreated, insomnia increases the risk of relapse and recurrence of depressive episodes, unintentional injuries, poor school performance, substance use, obesity, and the risk for suicide. This project seeks to develop a nonpharmacological treatment for insomnia in adolescents with depression that is feasible and effective. The specific methodologies that will help accomplish these results are: 1) use of focus groups of adolescents with depression and insomnia to determine how the current standard, nonpharmacological treatment for insomnia (cognitive-behavioral therapy for insomnia; CBTI) among adults can be modified for use by adolescents with depression and 2) determine the preliminary effectiveness, feasibility, and tolerability of group CBTI in adolescents with depression (CBTI-AD) developed using feedback from the focus groups. This project will help to improve the quality and scope of delivery of mental health services in Michigan by a) gaining a greater understanding of how sleep disturbance may perpetuate depression in adolescents and b) to provide mental health professionals with a nonpharmacological treatment option for insomnia in adolescents with depression.

ELIGIBILITY:
Inclusion Criteria:

* Between 13-19 years of age
* Are depressed
* Have insomnia

Exclusion Criteria:

* Are not depressed
* Do not have insomnia
* Currently using a sleep aid
* Have bipolar depression
* Have psychotic disorder
* Have a sleep disorder other than insomnia

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Change from baseline in insomnia at 5 weeks
  A 5-item insomnia severity questionnaire
Multidimensional Fatigue Inventory | Change from baseline in fatigue at 5 weeks
  A 14-item questionnaire on fatigue
Quick Inventory of Depressive Symptomatology | Change from baseline in depression at 5 weeks
  A 16-item questionnaire on depression

SECONDARY OUTCOMES:
Alcohol and drug use screening test (CRAFFT) | Baseline
  A six item questionnaire that assesses risk and substance use. This questionaire is delivered once at baseline.
Morningness Eveningness Questionnaire -modified | Baseline
  A 10 item questionnaire assessing phase preference of evening, morning, or neither; This questionaire is delivered once at baseline.

OTHER OUTCOMES:
Sleep diaries | Change from baseline in sleep at 5 weeks
  A subjective assessment of daily patterns of sleep

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States